CLINICAL TRIAL: NCT03305276
Title: Evaluation of the Impact of Mediterranean Lifestyle and Diet on Intermediate and Final Endpoints of Health
Brief Title: Observatory on Impact of Life Styles on Health Outcomes
Acronym: OIVITA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guido Iaccarino (Other)
Responsible Party: Sponsor-Investigator, Guido Iaccarino, Associate Professor of Internal Medicine, Azienda Ospedaliera OO.RR. S. Giovanni di Dio e Ruggi D'Aragona
Organization: Azienda Ospedaliera OO.RR. S. Giovanni di Dio e Ruggi D'Aragona (Other)
Other Study IDs: 1234
Record Dates: First submitted 2017-07-06; First posted 2017-10-09 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Outcome
Keywords: diet;; exercise;; hypertension;; vitamin d
MeSH Terms: conditions — Motor Activity; Hypertension

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- general population: the study is open to all population, (14-90 years, male/female) to verify the impact of lifestyles (mediterranean style) on intermediate and hard endpoint.

SUMMARY:
The present is an observational study conducted on the general population in villages of Southern Italy every year during the world hypertension day. So far, A total of 412 persons (193 males and 219 female, 14-85 years) were recruited during the XI and XII World Hypertension Day (2015 and 2016). The study was approved by the relevant institutional Ethical Committee of Salerno University.

DETAILED DESCRIPTION:
In occasion of the World Hypertension Day in may , boots are organized in the major squares of the southern italy villages, and volunteers of the Medical School of Salerno collect through means of questionnaires, anamnestic data and dietary habits, and measure blood pressure after 5 minutes in the sitting position, 3 times with an interval of 2 minutes using validated, ESH approved electronic oscillometer (A100, Microlife, Italy), according to the ESC/ESH guidelines. Other questions regard previous cardiovascular conditions or events (coronary heart disease) and cardiovascular accidents (TIA and stroke). Eventual drug treatment and Vitamin D supplementation is also annotated. A venous blood sample is drawn from the antecubital vein and blood is stored for biochemical analysis at the University Hospital Centralized Service. Data are digitally stored for analysis.

Anamnestic and biochemical data regarding age, sex-specific cholesterol, HDL cholesterol, systolic BP and cigarette smoking pre-existing conditions and way of life are used for the calculation of cardiovascular risk according to the Framingham Cardiovascular Risk Score. Familiarity for cardiovascular disease is defined as cardiovascular events in parents and siblings less than 50 years old.

The validated questionnaire alternate Mediterranean Diet Score (aMed), is administered to assess adherence to the Mediterranean Diet . Laboratory assessment of blood samples. A venous blood sample was collected in two tubes of 5.0 ml and centrifuged in the day. The time of the last meal was recorded during the data collection. Blood glucose, insulin, blood urea nitrogen (BUN), creatinine, calcium, phosphorus, total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides, 25(OH)D, PTH, Vitamin B-12 and folic acid are assessed. Glomerular filtration rate (GFRs) is estimated using the equation of Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) .

ELIGIBILITY:
Inclusion Criteria:

- General population

Exclusion Criteria:

* Subjects who do not sign informed consent and do not give authorization will be excluded from the study
* Subjects fed through parenteral feeding

Ages: 14 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Volunteers from Southern Italy will be recruited in occasion of health promoting events in villages.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2014-05-16 (Actual); Primary Completion 2020-07-16 (Estimated); Study Completion 2024-05-16 (Estimated)

PRIMARY OUTCOMES:
cardiovascular events | 10 year
  Presence of events in the anamnesis of subjects enrolled

SECONDARY OUTCOMES:
cardiovascular risk | 10 years
  Framingham Risk Score

OTHER OUTCOMES:
vitamin D profile | 10 years
  vitamin d serum levels will be assessed and compared to the life style
vitamin B12 profile | 10 years
  vitamin b12 serum levels will be assessed and compared to the life style
Folic Acid profile | 10 years
  folic acid serum levels will be assessed and compared to the life style

CONTACTS AND LOCATIONS:
Locations (1):
- San Giovanni e Ruggi Hospital, Salerno, Italy

IPD SHARING:
Plan to Share IPD: No